CLINICAL TRIAL: NCT04896502
Title: Effectiveness of Telemedicine Home Assessments for Identification and Reduction of Asthma Triggers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 239759
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2023-03

CONDITIONS: Asthma in Children
Keywords: Asthma; Telemedicine
MeSH Terms: conditions — Asthma | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Arm (Experimental): For the proposed study, participants will randomized to receive TM home assessments/interventions performed by a trained home visitor (HV) or standard of care asthma trigger education by the HV. Those who are randomized to TM home assessments/interventions will complete a baseline home assessment and two follow-up visits, 2 months apart. Visits will assess the presence of potential asthma triggers in the home and frequency of asthma symptoms/exacerbations. TM participants will be provided education and materials necessary to reduce asthma triggers in the home. Follow-up visits will assess the interval change in presence of asthma triggers, change in daily asthma symptoms/exacerbations, and participant/family retention of education.
  Interventions: Other: Interactive Video (IAV) Telemedicine
- Standard of Care Education (Active Comparator): For subjects randomized to receive standard of care asthma education, written and verbal information will be provided regarding identification and removal of potential asthma triggers in the home but no formal assessment of the home will be performed, nor will participants in this arm receive trigger reduction materials.
  Interventions: Behavioral: Standard of Care Education

INTERVENTIONS:
Behavioral: Standard of Care Education — Education regarding recognition and removal of in-home asthma triggers
  Arms: Standard of Care Education
Other: Interactive Video (IAV) Telemedicine — Interactive video assessment of asthma triggers in the home.
  Arms: Telemedicine Arm

SUMMARY:
The study is about comparing asthma home assessments/interventions by telemedicine compared to providing education alone. Interactive Video (IAV) defines telemedicine. It allows two-way communication in real-time with both audio and visual communication between the subject and someone from the study team. It is similar to using Face Time on a mobile device. Asthma home assessments/interventions are used to identify things in a home that can make asthma symptoms worse, called triggers. Reducing these triggers in the home can improve asthma.

DETAILED DESCRIPTION:
In this study, supplies will be given to some participants to help reduce or remove triggers from the home. One example is dust mites. These are microscopic bugs that are found in every home, cannot be seen by the naked eye, and make asthma symptoms worse. Part of the study includes collecting two dust samples from home to check dust mite levels at the beginning of the study and at the end. This study may help elucidate whether telemedicine home assessments work better than education alone at lowering dust mite levels and improving a child's asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 5 years and ≤ 18 years
2. Have a diagnosis of persistent asthma as defined by national guidelines criteria1
3. Patient receives care in Arkansas Children's Hospital (ACH) primary care, in patient and/or specialty clinics
4. Patient has had at least one or more acute exacerbations of asthma within the 12 months prior to enrollment that led to an emergency department visit, hospital admission, or prescription for systemic steroids
5. English speaking participants/parents
6. Access to WIFI, smartphone or mobile device (tablet)

Exclusion Criteria:

1. Age <5 or >18 years
2. Non-English speaking participants/parents
3. Patients not receiving primary and/or asthma specialty care or inpatient services at ACH
4. Inability of patient or family to participate in TM evaluation due to lack of access to WIFI or smartphone or mobile device

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pesek, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telemedicine Arm | Standard of Care Education
Started | 13 | 14
Completed | 3 | 4
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemedicine Arm | Standard of Care Education | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 14 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.52 (3.27) | 8.76 (3.59) | 10.14 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 2 | 3 | 5
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Significant Change in D. Pteronyssinus Levels at End of Study Evaluation
Description: Comparison of D. pteronyssinus levels collected in participant homes at baseline and at end of study with measure of number of subjects with a significant change
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Arm | Standard of Care Education
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

2. Secondary Outcome: Differences in ACT Score Between Telemedicine and Standard of Care Groups
Description: We will measure differences in ACT scores from baseline to 6 months between the Telemedicine and Standard of Care groups. Asthma Control Test (ACT) is a 5 question (<12 years of age) or 7 question (>/= 12 years of age) test utilized to assess asthma control. Scores range from 0 to 25. The maximum score is 25 and a score of 19 or less indicates "not well-controlled" asthma.
Time Frame: 6 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Telemedicine Arm | Standard of Care Education
Number analyzed (Participants) | 3 | 4
score on a scale
  Enrollment ACT score | 23.3 (2.36) | 21.25 (2.165)
  6 Month ACT score | 23.3 (2.36) | 22 (3)

3. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction measured by standardized survey. Respondents were asked "How satisfied were you with your overall experience?" and were scored on a scale from "Complete Satisfied" to "Not at All Satisfied"
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Telemedicine Group: For the proposed study, participants will randomized to receive TM home assessments/interventions performed by a trained home visitor (HV) or standard of care asthma trigger education by the HV. Those who are randomized to TM home assessments/interventions will complete a baseline home assessment and two follow-up visits, 2 months apart. Visits will assess the presence of potential asthma triggers in the home and frequency of asthma symptoms/exacerbations. TM participants will be provided education and materials necessary to reduce asthma triggers in the home. Follow-up visits will assess the interval change in presence of asthma triggers, change in daily asthma symptoms/exacerbations, and participant/family retention of education.
  Interactive Video (IAV) Telemedicine: Interactive video assessment of asthma triggers in the home.
Arm/Group | Telemedicine Group | Standard of Care Education
Number analyzed (Participants) | 8 | 9
Participants
  Completely satisfied | 4 | 4
  Very satisfied | 2 | 1
  Somewhat satisfied | 0 | 0
  Not at all satisfied | 0 | 0
  Missing data | 2 | 4

ADVERSE EVENTS:
Time Frame: 6 months
Description: No patients experienced an adverse event, serious adverse event, or mortality during the study period
Arm/Group | Telemedicine Arm | Standard of Care Education
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT04896502/Prot_SAP_000.pdf